CLINICAL TRIAL: NCT05649813
Title: Prospective Registry on Chronic RhinoSinusitis With Nasal Polyps In the Greater Gulf Region
Brief Title: A Study in Male and Female Adult Participants With Chronic Rhinosinusitis With Nasal Polyps In the Greater Gulf Region
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17627; U1111-1279-3286 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-11-15; First posted 2022-12-14 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRSwNP: Participants with CRSwNP in the Gulf region

SUMMARY:
Primary Objective:

- To describe the clinical characteristics of participants with chronic rhinosinusitis with nasal polyps (CRSwNP) in terms of disease severity, Type 2 inflammation-related comorbidities (such as asthma and allergic rhinitis), other associated comorbidities, and treatments used in a real-world setting

Secondary Objectives:

* Describe the progression in treatment outcomes at different visits (baseline, 3 months, 6 months, and 12 months).
* To assess the healthcare resource utilization of participants with CRSwNP in countries of the Gulf region (number of visits, emergency room (ER), surgery, etc).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants.
* Participants diagnosed with chronic rhinosinusitis with nasal polyps (CRSwNP) for at least one year prior to study start.
* Participants diagnosed with CRSwNP according to criteria of American Academy of Otolaryngology-Head and Neck Surgery (i.e. the diagnosis is confirmed in medical records by clinical symptoms and objective evidence of nasal polyps by using anterior rhinoscopy and nasal endoscopy when available and/or computed tomography (CT) scan).
* Participants should be at least 18 years old.
* Participants must have signed an informed consent.

Exclusion Criteria:

* Participants with chronic rhinosinusitis without nasal polyps (CRSsNP)
* Pregnant/breastfeeding participants or participants planning for a pregnancy.
* Participants participating in other interventional clinical trials involving any investigational drug.
* Participants with granulomatous diseases such as vasculitis or sarcoidosis. The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CRSwNP
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with mild, moderate or severe disease (measured by visual analogue scale [VAS] score) | Day 0 (baseline) to Month 12
The mean baseline Sinonasal Outcome Test (SNOT-22) scores | Day 0
The mean baseline nasal polyps score (NPS) | Day 0
Percentage of participants with Type 2 inflammation-related comorbidities including bronchial asthma, allergic rhinitis, atopic dermatitis, chronic spontaneous urticaria, eosinophilic esophagitis (EoE), and food allergy | Day 0
Percentage of participants with other associated comorbidities including chronic obstructive pulmonary disease (COPD), ulcerative colitis, eosinophilic gastritis, or other comorbidities (if relevant) | Day 0
Percentage of different medications used by participants with CRSwNP during the follow-up period as per decision of the treating physician | Day 0 to Month 12

SECONDARY OUTCOMES:
The mean change in the baseline Sinonasal Outcome Test (SNOT-22) scores | Day 0 (baseline), Month 3, Month 6, and Month 12
The mean change in the baseline nasal polyps score (NPS) | Day 0, Month 3, Month 6, and Month 12
Mean change in the baseline total symptoms score (TSS) | Day 0, Month 6, and Month 12
The proportion of CRSwNP patients with hospitalization | Day 0 to Month 12
The proportion of CRSwNP patients with emergency room (ER), office, or general practitioner visits | Day 0 to Month 12
The mean number of days/visits to ER, office, or general practitioner | Day 0 to Month 12
The mean number of days of sick leaves | Day 0 to Month 12
The proportion of surgical procedures performed during the hospital visit including nasal polypectomy with additional sinus dissection, isolated nasal polypectomy, or functional endoscopic sinus surgery [FESS]) | Day 0 to Month 12
The mean number of participants with CRSwNP who need surgical treatment | Day 0 to Month 12
Total number of surgeries | Day 0 to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number: 01, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org